CLINICAL TRIAL: NCT01035788
Title: Effects of Mindfulness-Based Cognitive-Behavioral Conjoint Therapy on PTSD and Relationship Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B7331-R; 1001-02B (Other: IUPUI IRB)
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: PTSD
Keywords: PTSD; mindfulness meditation; cognitive behavior therapy; relationship function; couple therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based CBCT (Experimental): Mindfulness Based Cognitive Behavioral Conjoint Therapy for PTSD
  Interventions: Behavioral: Mindfulness Based Cognitive Behavioral Conjoint Therapy
- CBCT Communication Skills (Active Comparator): CBCT for PTSD - Communication Skills
  Interventions: Behavioral: CBCT for PTSD - Communication Skills

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Behavioral Conjoint Therapy — This intervention combines Cognitive Behavioral Conjoint Therapy for PTSD and mindfulness skills. Cognitive Behavioral Conjoint Therapy for PTSD includes PTSD psychoeducation, communication skills training and cognitive restructuring. Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses.
  Arms: Mindfulness-Based CBCT
Behavioral: CBCT for PTSD - Communication Skills — This control intervention will provide psychoeducation including the communication skills content from sessions 1-7 of Cognitive Behavioral Conjoint Therapy for PTSD.
  Arms: CBCT Communication Skills

SUMMARY:
The purpose of this study is to first adapt Cognitive Behavioral Conjoint Therapy for PTSD for Operation Enduring Freedom and Operation Iraqi Freedom (OEF-OIF) Veterans diagnosed with PTSD and their intimate partners by (1) reducing the overall length of treatment from 15 weeks to 10 weeks through the use of a weekend couple retreat to deliver the first two of three phases of the three-phase protocol; and (2) by integrating mindfulness interventions as a way to mitigate the short, more condensed treatment. Secondly, this study will examine the effects of this adapted Mindfulness-Based Cognitive-Behavioral Conjoint Therapy on PTSD symptoms and intimate relationship functioning.

DETAILED DESCRIPTION:
Between 5 and 15 percent of Veterans return from deployment in Iraq and Afghanistan with PTSD and the symptoms adversely affect many aspects of their lives, including intimate relationships. Although research findings consistently suggest that the degree of intimate relationship dysfunction correlates with the severity of Veteran's PTSD symptoms, few couples interventions have been developed and systematically evaluated. Cognitive Behavioral Conjoint Therapy for PTSD (CBCT for PTSD) is an intervention developed to treat both PTSD and relationship dysfunction that has shown promising preliminary results. However, the literature suggests that OEF-OIF Veterans prefer shorter time-limited treatments and CBCT for PTSD requires as many as 15 sessions. CBCT for PTSD lacks specific interventions that train meta-awareness, such as those taught in mindfulness-based stress reduction (MBSR). Mindfulness practices have an emerging evidence base for improving both PTSD and relationship functioning in several important ways. First, practicing mindfulness promotes the relaxation response which counters hyperarousal and results in a calmer approach to difficulties and challenges. Second, avoidance and numbing are countered by mindfully allowing one's experience to be as it is while suspending judgment, which is associated with increased compassion and empathy. Lastly, mindfulness supports a way of being with all life experiences rather than providing techniques just for coping with specific difficulties, which enables individuals to access inner strengths that are already available to them. Just as many physical conditions require more than one rehabilitation approach, there may be a synergy between CBCT for PTSD and mindfulness interventions. Mindfulness skills may assist individuals in tolerating painful emotional reactions to their experiences which may in turn enhance their awareness of associated feelings and thoughts. With enhanced meta-awareness the beliefs that may maintain PTSD symptoms and relationship dysfunction become more amenable to cognitive restructuring. Therefore, the goal of this study is to examine the effects of a Mindfulness-Based adaptation of CBCT for PTSD. The study involves two phases over the course of four years. In Phase 1, mindfulness interventions will be integrated within the Cognitive Behavioral Conjoint Therapy for PTSD treatment manual and the content of the first 7 sessions of CBCT will be adapted to be delivered during a weekend retreat. The integrated intervention, MB-CBCT for PTSD, will be delivered to 10 OIF-OEF Veterans and each of their intimate partners in order to develop and test procedures to train and monitor therapists. During Phase 2, 40 OEF-OIF Veterans and each of their intimate partners will be consented and a randomized controlled trial with be conducted comparing the MB-CBCT for PTSD with a control condition that teaches communication skills drawn from the first 7 sessions of the CBCT manual. We hypothesize that MB-CBCT for PTSD will lead to greater improvement in: 1) Veterans' PTSD symptoms as measured by the Clinician Administered PTSD Scale (primary outcome) and PTSD Checklist (secondary outcome); 2) Veterans' and partners' relationship functioning (secondary outcome); and 3) anxiety and depression symptoms (secondary outcomes). PTSD constitutes a substantial proportion of the burden of illness among Veterans. The longer term goals of this project are to conduct a fully-powered randomized controlled clinical trial of MB-CBCT to determine its effectiveness and to finalize the treatment manual.

ELIGIBILITY:
Inclusion Criteria:

Veteran must:

* be enrolled in outpatient treatment
* have a confirmed diagnosis of PTSD
* have no major change in psychiatric medication for at least 1 month
* have a partner mutually committed to maintaining the relationship for the duration of the intervention
* willing to forgo initiating psychotherapy for PTSD or other conditions during the study

Exclusion Criteria:

* severe physical or sexual relationship aggression in the past year
* current suicidal/homicidal intent (Veteran or partner)
* cognitive impairment that precludes understanding session content (either Veteran or partner)
* current substance dependence of Veteran or partner
* uncontrolled psychotic or bipolar disorder in Veteran or partner
* PTSD diagnosis in the partner
* self-mutilation or self-injury within the previous 6 months by Veteran or partner
* unwilling to have therapy or CAPS sessions video or audio recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louanne Whitman Davis, PsyD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 88 couples (88 Veterans & their 88 intimate partners) were consented & 78 couples completed eligibility screening. 32 couples were excluded (not meeting inclusion/exclusion criteria; met criteria but declined to proceed, or unable to attend required retreat weekend. The remaining 46 couples were randomized (46 Veterans & 46 partners).
Groups:
- Mindfulness-Based Cognitive-Behavioral Conjoint Therapy: Mindfulness-Based Cognitive-Behavioral Conjoint Therapy for PTSD (MB-CBCT) is an adaptation of Cognitive-Behavioral Conjoint Therapy for PTSD (CBCT) that offers CBCT Phases 1 and 2 plus mindfulness training in a couple weekend retreat format, followed by continued use of mindfulness skills in session and for out of session practice during one transition couple therapy session, followed by CBCT Phase 3 couple sessions.
- Cognitive Behavioral Conjoint Therapy Communication Skills: Cognitive-Behavioral Conjoint Therapy (CBCT) phases 1-2 communications skills training (no PTSD psychoeducation) offered during a weekend couple retreat followed by two monthly group couple sessions for skills review.
Period: Overall Study
Arm/Group | Mindfulness-Based Cognitive-Behavioral Conjoint Therapy | Cognitive Behavioral Conjoint Therapy Communication Skills
Started | 23 (23 couples = 23 Veterans + 23 partners; only data for Veterans will be included for primary outcome.) | 23 (23 couples = 23 Veterans + 23 partners; only data for Veterans will be included for primary outcome.)
Completed | 17 | 9
Not Completed | 6 | 14

BASELINE CHARACTERISTICS:
Population: Data is included for Veterans only since this was the data needed for the primary outcome analysis of the Clinician Administered PTSD Scale for the Veteran participants who had PTSD.
Groups:
- Mindfulness-Based Cognitive-Behavioral Conjoint Therapy: Mindfulness Based Cognitive Behavioral Conjoint Therapy for PTSD
  Mindfulness Based Cognitive Behavioral Conjoint Therapy for PTSD: This intervention combines cognitive behavioral conjoint therapy for PTSD and mindfulness skills. Cognitive behavioral conjoint therapy for PTSD includes psychoeducation, skills training and cognitive restructuring. Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses.
- Cognitive Behavioral Conjoint Therapy Communication Skills: Psychoeducational Intervention
  Psychoeducation (control): This control intervention will provide psychoeducation including the communication content from sessions 1-7 of cognitive behavioral conjoint therapy for PTSD.
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Cognitive-Behavioral Conjoint Therapy | Cognitive Behavioral Conjoint Therapy Communication Skills | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (9.2) | 41.0 (11.3) | 39.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 22 | 19 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Clinician Administered PTSD Scale (CAPS) [Mean (Standard Deviation); unit: units on a scale] — The Clinician Administered PTSD Scale (CAPS) is a semi-structured interview that evaluates PTSD symptoms and diagnostic status according to the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (APA, 2000). The intensity and frequency of each symptom is separately on a 5 point Likert scale ranging from zero to four. The total CAPS symptom severity score ranges from 0-136, with higher scores indicating greater PTSD symptoms severity. For the purposes of this study, a score of 45 or greater confirmed a diagnosis of PTSD.
  units on a scale | 71.1 (12.4) | 70.4 (13.9) | 70.7 (13.1)
PTSD Checklist (PCL) [Mean (Standard Deviation); unit: units on a scale] — The PTSD Checklist (PCL) is a 17-item self-report measure of PTSD symptom severity corresponding to the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (APA, 2000) PTSD symptoms. The score range is 17-85 and higher scores indicated greater PTSD symptoms severity.
  units on a scale | 57.6 (7.8) | 57.2 (10.5) | 57.4 (9.2)
Dyadic Adjustment Scale (DAS) [Mean (Standard Deviation); unit: units on a scale] — The Dyadic Adjustment Scale (DAS) is a 32-item self-report inventory designed to measure partner perceptions of the quality of an intimate dyadic relationship. Scores range from 0-151, with higher scores indicating higher satisfaction. A total score of 98 or higher indicates relationship satisfaction.
  units on a scale | 99.7 (19.2) | 96.0 (25.0) | 97.9 (22.1)
Beck Depression Inventory II (BDI) [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI) is a 21 item self-report measure of symptoms of depression over the course of the past two weeks. Items are rated on a 4-point scale ranging from zero to three. Ratings for each item are summed yielding total scores between zero and 63. Higher scores indicate higher levels of depressive symptoms.
  units on a scale | 25.6 (9.5) | 26.8 (9.6) | 26.2 (9.5)
State-Trait Anxiety Inventory State Subscale [Mean (Standard Deviation); unit: units on a scale] — The State subscale of the State-Trait Anxiety Inventory (STAI) is a self-report measure of current anxiety symptoms. The scores range 20-80 and higher scores indicate higher levels of current anxiety.
  units on a scale | 51.9 (8.3) | 49.8 (12.7) | 50.9 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: The Clinician Administered PTSD Scale (CAPS; Blake et al., 1995) is a semi-structured interview that evaluates PTSD symptoms and diagnostic status according to the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (APA, 2000). The intensity and frequency of each symptom is separately on a 5 point Likert scale ranging from zero to four. The total CAPS symptom severity score ranges from 0-136, with higher scores indicating greater PTSD symptoms severity. For the purposes of this study, a score of 45 or greater confirmed a diagnosis of PTSD.
Time Frame: treatment end (approximately 10 weeks after session 1 of the interventions)
Population: This analysis was intention to treat and included the 30 participants of the original 34 who completed the CAPS interview at treatment end.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mindfulness-Based Cognitive-Behavioral Conjoint Therapy: Mindfulness Based Cognitive Behavioral Conjoint Therapy for PTSD
  This intervention combines cognitive behavioral conjoint therapy for PTSD and mindfulness skills. Cognitive Behavioral ConjointTtherapy for PTSD includes psychoeducation, skills training and cognitive restructuring. Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses.
- Cognitive Behavioral Conjoint Therapy Communication Skills: Cognitive-Behavioral Conjoint Therapy for PTSD - Communication Skills
  This control intervention will provide communication skills training from sessions 1-7 of Cognitive Behavioral Conjoint Therapy for PTSD.
Arm/Group | Mindfulness-Based Cognitive-Behavioral Conjoint Therapy | Cognitive Behavioral Conjoint Therapy Communication Skills
Number analyzed (Participants) | 19 | 11
units on a scale | 45.5 [36.6 to 54.5] | 46.2 [34.9 to 57.5]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive-Behavioral Conjoint Therapy vs Cognitive Behavioral Conjoint Therapy Communication Skills; We sought to obtain a sample size of 18 per group to provide 80% power to detect a .97 standard deviation difference in mean change in CAPS between MB-CBCT and the CBCT-Communication Skills at treatment end based on a two-tailed t-test at 5% significance. Linear mixed models with repeated measures were performed to address the primary hypotheses that MB-CBCT would result in a greater improvement for Veterans and their partners than CBCT-Communication Skills at the end of treatment; Test type: Superiority or Other; p = .849, Mixed Models Analysis; p value was obtained from the contrast of the linear mixed model; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-1.39 to 13.2], Standard Error of Mean 7.24

ADVERSE EVENTS:
Time Frame: 4 years
Description: Adverse events were assessed for both veterans and their partners separately. There were no adverse events for veterans or their partners.
Groups:
- Mindfulness-Based Cognitive-Behavioral Conjoint Therapy: Mindfulness Based Cognitive Behavioral Conjoint Therapy for PTSD
  Mindfulness Based Cognitive Behavioral Conjoint Therapy: This intervention combines Cognitive Behavioral Conjoint Therapy for PTSD and mindfulness skills. Cognitive Behavioral Conjoint Therapy for PTSD includes PTSD psychoeducation, communication skills training and cognitive restructuring. Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses.
- Cognitive Behavioral Conjoint Therapy Communication Skills: CBCT for PTSD - Communication Skills
  CBCT for PTSD - Communication Skills: This control intervention will provide psychoeducation including the communication skills content from sessions 1-7 of Cognitive Behavioral Conjoint Therapy for PTSD.
Arm/Group | Mindfulness-Based Cognitive-Behavioral Conjoint Therapy | Cognitive Behavioral Conjoint Therapy Communication Skills
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

LIMITATIONS AND CAVEATS:
Detecting significant differences between groups may be limited by loss to follow-up of 3x more CBCT-S subjects than MB-CBCT. Differences between CAPS and PCL ratings may suggest issues with CAPS assessors although inter-rater reliability was strong.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes